CLINICAL TRIAL: NCT03952559
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Outpatient Study Evaluating the Pharmacokinetics, Efficacy, and Safety of Baricitinib in Pediatric Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Baricitinib (LY3009104) in Children and Adolescents With Atopic Dermatitis
Acronym: BREEZE-AD-PEDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16966; I4V-MC-JAIP (Other: Eli Lilly and Company); 2018-000349-38 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants were randomized to one of the four double-blind treatment arms. A separate group of 33 participants received open label baricitinib as part of pharmacokinetic (PK) lead-in (not randomized) period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Baricitinib Open Label High Dose (PK Lead-in) (Experimental): Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension (1 mL) QD.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid
- Baricitinib High Dose (Experimental): Participants 10 to < 18 years received Baricitinib high dose (4 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid
- Baricitinib Medium Dose (Experimental): Participants 10 to < 18 years received Baricitinib low dose (1 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib low dose (0.5 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid
- Baricitinib Low Dose (Experimental): Participants 10 to < 18 years received Baricitinib low dose (1 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib low dose (0.5 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Topical corticosteroid
- Placebo (Placebo Comparator): Participants 10 to < 18 years received placebo tablets. Participants 2 to < 10 years received placebo as oral suspension.
  Interventions: Drug: Placebo; Drug: Topical corticosteroid

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib High Dose; Baricitinib Low Dose; Baricitinib Medium Dose; Baricitinib Open Label High Dose (PK Lead-in)
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Topical corticosteroid — Administered as standard-of-care

SUMMARY:
The reason for this study is to see if the study drug called baricitinib works and is safe in children and teenage participants with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* At or above the 5th percentile of weight for age.
* Have been diagnosed with moderate to severe atopic dermatitis for at least 12 months (if 6 years old or older) or at least 6 months (if 2 up to 6 years old).
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episode of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to beginning study treatment.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor.
  * Received any parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned initiation of study drug or are anticipated to require parenteral injection of corticosteroids during the study.
* Have had an intra-articular corticosteroid injection within 2 weeks prior to study entry or within 6 weeks prior to planned initiation of study drug.
* Have high blood pressure characterized by a repeated systolic or diastolic blood pressure >95th percentile based on age, sex and height.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster (shingles or chicken pox), tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 516 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (78):
- Argentina (4):
  - Instituto de Neumonología Y Dermatología, Capital Federal, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundacion CIDEA, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundación Respirar, Buenos Aires
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Wien, Vienna, Vienna
  - Sozialmedizinisches Zentrum Ost/Donauspital, Vienna, Vienna
- Brazil (5):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - IDERJ - Instituto de Dermatologia e Estética do Brasil, Rio de Janeiro
  - Hospital do Servidor Público Estadual - IAMSPE - centro de estudos urológicos, São Paulo
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín, Nový Jičín
  - Fakultni Nemocnice v Motol, Prague, Praha 5
  - Fakultni nemocnice Bulovka, Prague, Praha 8
  - Sanatorium profesora Arenbergera, Prague
- France (7):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice, Alpes-Maritimes
  - Hôpitaux Drôme Nord - Romans, Romans-sur-Isère, Drôme
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Finistère
  - Hôpital Saint Vincent de Paul, Lille, Hauts-de-France
  - Chu Saint Eloi, Montpellier, Languedoc-Roussillon
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Loire-Atlantique
  - CHU de Toulouse - Hopital Larrey, Toulouse, Midi-Pyrénées
- Germany (4):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Katholisches Kinderkrankenhaus Wilhelmstift, Hamburg
- Hungary (2):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
- India (3):
  - B. J. Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Aakash Healthcare: Super Speciality Hospital -Dwarka, Dwarka, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
- Israel (4):
  - Sheba Medical Center, Ramat Gan, Central District
  - Emek Medical Center, Afula, Northern District
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Japan (10):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Takeda Dermatology Skincare Clinic, Sapporo, Hokkaido
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - National Mie Hospital, Tsu, Mie-ken
  - Kume Clinic, Sakai, Osaka
  - Senri-Chuo Hanafusa Dermatology Clinic, Toyonaka, Osaka
  - Dokkyo Medical University Hospital, Shimotsuga, Tochigi
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
  - Shinjuku Minamiguchi Hifuka, Tokyo
- Mexico (5):
  - Centro de Atención en Enfermedades Inflamatorias CATEI, Guadalajara, Jalisco
  - Centro Regiomontano de Investigación, Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Arké SMO S.A de C.V, Veracruz
- Poland (3):
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Specjalistyczne Gabinety Lekarskie "DERMED" Anna Kaszuba, Lodz, Łódź Voivodeship
- Russia (4):
  - Krasnodar Clinical Skin and Venereal Diseases Dispensary, Krasnodar, Krasnodarskiy Kray
  - Children's Health Research Center of RAMS, Moscow, Moscow
  - Moscow Scientific and Practical Center of Dermatovenerology and Cosmetology - Central branch, Moscow, Moscow
  - Tula Regional Clinical Dermatovenerological Dispensary, Tula, Tula Oblast
- Spain (7):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona [Barcelona]
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CHOP-Centro De Especialidades De Mollabao, Pontevedra, Pontevedra [Pontevedra]
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (6):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- United Kingdom (3):
  - Royal Hospital for Sick Children, Glasgow, Glasgow City
  - St Thomas's Hospital, London, London, City of
  - Queen's Medical Centre, Nottingham University Hospitals, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wollenberg A, Ikeda M, Chu CY, Eichenfield LF, Seyger MMB, Prakash A, Angle R, Zhu D, Pontes M, Paller AS. Longer-term safety and efficacy of baricitinib for atopic dermatitis in pediatric patients 2 to <18 years old: a randomized clinical trial of extended treatment to 3.6 years. J Dermatolog Treat. 2024 Dec;35(1):2411834. doi: 10.1080/09546634.2024.2411834. Epub 2024 Nov 10. PMID 39522957
- See also: A Study of Baricitinib (LY3009104) in Children and Adolescents With Atopic Dermatitis (BREEZE-AD-PEDS) — https://trials.lillytrialguide.com/en-US/trial/B796sBY99npuSW6LYeHAk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 516 participants (33+483=516) were enrolled in the study. Of which 483 participants were randomized to one of the four double-blind treatment arms, and 33 participants received open label baricitinib as part of pharmacokinetics (PK) lead-in (not randomized).
Groups:
- Baricitinib Open Label High Dose (PK Lead-in): Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Placebo Double-blind: Participants 10 to < 18 years received placebo tablets. Participants 2 to < 10 years received placebo as oral suspension.
- Baricitinib Double-blind Low Dose: Participants 10 to < 18 years received Baricitinib low dose (1 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib low dose (0.5 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
- Baricitinib Double-blind Medium Dose: Participants 10 to < 18 years received Baricitinib medium dose (2 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib medium dose (1 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
- Baricitinib Double-blind High Dose: Participants 10 to < 18 years received Baricitinib high dose (4 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
Period: High Dose Open Label - PK Lead-in
Arm/Group | Baricitinib Open Label High Dose (PK Lead-in) | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Started | 33 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 33 | 0 | 0 | 0 | 0
Completed | 33 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Double Blind Treatment Period
Arm/Group | Baricitinib Open Label High Dose (PK Lead-in) | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Started | 0 (Participants who completed the Open-label PK Lead-in (Week 2) continued into the long-term extension study.) | 122 (Participants were assigned to this arm during double blind treatment period.) | 121 (Participants were assigned to this arm during double blind treatment period.) | 120 (Participants were assigned to this arm during double blind treatment period.) | 120 (Participants were assigned to this arm during double blind treatment period.)
Received at Least One Dose of Study Drug | 0 | 122 | 120 | 120 | 120
Completed | 0 | 115 | 116 | 117 | 119
Not Completed | 0 | 7 | 5 | 3 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 4 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2 | 0
Not completed — Inadvertently randomized | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug in the PK Lead-in period (Study period 1).
  All randomized participants in the double-blind treatment period (Study period 2).
Groups:
- Baricitinib Open Label High Dose: Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Total: Total of all reporting groups
Arm/Group | Baricitinib Open Label High Dose | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose | Total
Number analyzed (Participants) | 33 | 122 | 121 | 120 | 120 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.28 (4.296) | 11.75 (4.012) | 12.35 (4.052) | 11.81 (3.661) | 11.93 (3.829) | 11.92 (3.914)
Age, Customized [Count of Participants; unit: Participants]
  2 to <6 years | 6 | 14 | 9 | 8 | 9 | 46
  6 to <10 years | 7 | 20 | 24 | 26 | 23 | 100
  10 to <18 years | 20 | 88 | 88 | 86 | 88 | 370
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 64 | 62 | 63 | 53 | 262
  Male | 13 | 58 | 59 | 57 | 67 | 254
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 1 | 3 | 9
  Asian | 19 | 16 | 18 | 18 | 21 | 92
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5 | 4 | 14
  White | 13 | 94 | 94 | 93 | 88 | 382
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 8 | 4 | 2 | 4 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 0 | 16 | 18 | 18 | 18 | 70
  Hungary | 0 | 4 | 5 | 2 | 2 | 13
  Czechia | 0 | 6 | 7 | 4 | 5 | 22
  Japan | 0 | 9 | 10 | 10 | 9 | 38
  United Kingdom | 3 | 2 | 1 | 3 | 0 | 9
  India | 0 | 1 | 1 | 2 | 1 | 5
  Russia | 0 | 12 | 13 | 11 | 9 | 45
  Spain | 10 | 7 | 6 | 6 | 7 | 36
  Austria | 0 | 1 | 3 | 1 | 2 | 7
  Taiwan | 18 | 5 | 4 | 3 | 11 | 41
  Brazil | 0 | 7 | 9 | 7 | 11 | 34
  Poland | 0 | 19 | 19 | 25 | 26 | 89
  Mexico | 0 | 13 | 7 | 7 | 7 | 34
  Israel | 2 | 8 | 11 | 10 | 8 | 39
  Australia | 0 | 3 | 1 | 6 | 0 | 10
  France | 0 | 8 | 4 | 2 | 4 | 18
  Germany | 0 | 1 | 2 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥2 Point Improvement
Description: Percentage of participants achieving IGA of 0 or 1 with a ≥2 point improvement is presented. The IGA measures the investigator's global assessment of the participant's overall severity of their Atopic Dermatitis, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 16.4 | 18.2 | 25.8 | 41.7
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.7261, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.58 to 2.21]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.0718, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.95 to 3.41]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.73, 95% CI 2-sided [2.02 to 6.89]

2. Primary Outcome: Open Label Population Pharmacokinetics (Pop PK): Maximum Observed Drug Concentration at Steady State (Cmax,ss) of LY3009104
Description: Open label Pop PK: Cmax,ss was derived by a population pharmacokinetics approach.
Time Frame: Predose; 0.25 hours (h); 0.5 h; 1 h; 2-4 h; 4 h and 4-6 h post dose
Population: All participants who received at least one dose of study drug in the PK Lead-in (PK LI) period and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Baricitinib Open Label High Dose 2 to <6: Participants 2 to < 6 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Baricitinib Open Label High Dose 6 to <10: Participants 6 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Baricitinib Open Label High Dose 10 to <18: Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
Arm/Group | Baricitinib Open Label High Dose 2 to <6 | Baricitinib Open Label High Dose 6 to <10 | Baricitinib Open Label High Dose 10 to <18
Number analyzed (Participants) | 6 | 7 | 20
nanogram per milliliter (ng/mL) | 63.2 (30) | 40.1 (32) | 50.6 (29)

3. Primary Outcome: Open Label Pop PK: Area Under the Concentration-Time Curve for Dosing Interval at Steady State (AUCtau,ss) of LY3009104
Description: Open label Pop PK: AUCtau,ss was derived by a population pharmacokinetics approach.
Time Frame: Predose; 0.25 h; 0.5 h; 1 h; 2-4 h; 4 h and 4-6 h post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Baricitinib Open Label High Dose 10 to <18: Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally QD.
Arm/Group | Baricitinib Open Label High Dose 2 to <6 | Baricitinib Open Label High Dose 6 to <10 | Baricitinib Open Label High Dose 10 to <18
Number analyzed (Participants) | 6 | 7 | 20
hour*nanogram per milliliter (h*ng/mL) | 251 (18) | 178 (18) | 290 (44)

4. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
  The results were analyzed using non-responder imputation (NRI). All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as EASI75.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 32 | 32.2 | 40 | 52.5
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.9615, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.59 to 1.74]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.2010, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.83 to 2.41]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0017, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.38 to 3.95]

5. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
  The results were analyzed using non-responder imputation (NRI). All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as EASI90.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 12.3 | 11.6 | 21.7 | 30.0
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.8544, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.43 to 2.01]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.0561, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.98 to 3.91]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.54 to 5.82]

6. Secondary Outcome: Change From Baseline in EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs (1) erythema (2)edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score is obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Square (LS) Means were calculated using a mixed model repeated measures (MMRM) model with treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants in the double-blind treatment period and had evaluable EASI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 105 | 109 | 113 | 115
units on a scale | -14.16 (1.001) | -15.67 (0.990) | -15.83 (0.978) | -16.88 (0.984)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.2627, Mixed Models Analysis; LS Mean difference (Final Values) = -1.51, 95% CI 2-sided [-4.16 to 1.14], Standard Error of Mean 1.349
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.2135, Mixed Models Analysis; LS Mean difference (Final Values) = -1.67, 95% CI 2-sided [-4.31 to 0.97], Standard Error of Mean 1.342
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0443, Mixed Models Analysis; LS Mean difference (Final Values) = -2.72, 95% CI 2-sided [-5.36 to -0.07], Standard Error of Mean 1.347

7. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with visual analog scale (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 9.8 | 7.4 | 15.8 | 20.0
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.4943, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.30 to 1.78]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.1677, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.80 to 3.70]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0336, Regression, Logistic; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.06 to 4.70]

8. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement in Itch Numeric Rating Scale (NRS) for Participants 10 to <18 Years Old at Study Entry
Description: The Itch Numeric Rating Scale (NRS) is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participants itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 16
Population: All randomized participants (≥10 to <18 years old) in the double-blind treatment period and with baseline itch score >= 4.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Double-blind: Participants 10 to < 18 years received placebo tablets.
- Baricitinib Double-blind Low Dose: Participants 10 to < 18 years received Baricitinib low dose (1 mg) and placebo to maintain the blind, administered orally in tablet form QD.
- Baricitinib Double-blind Medium Dose: Participants 10 to < 18 years received Baricitinib medium dose (2 mg) and placebo to maintain the blind, administered orally in tablet form QD.
- Baricitinib Double-blind High Dose: Participants 10 to < 18 years received Baricitinib high dose (4 mg) and placebo to maintain the blind, administered orally in tablet form QD.
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 55 | 63 | 62 | 62
Percentage of participants | 16.4 | 17.5 | 25.8 | 35.5
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.8866, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.42 to 2.77]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.2316, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.70 to 4.26]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0328, Regression, Logistic; Odds Ratio, log = 2.59, 95% CI 2-sided [1.08 to 6.22]

9. Secondary Outcome: Percentage of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI50 is defined as a ≥ 50% improvement from baseline in EASI score.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 55.7 | 59.5 | 60.8 | 71.7
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.5361, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.70 to 1.98]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.4417, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.73 to 2.06]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0121, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.16 to 3.43]

10. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 4.1 | 5.0 | 5.0 | 12.5
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.7706, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.37 to 3.78]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.7409, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.38 to 3.86]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0253, Regression, Logistic; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.15 to 8.63]

11. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants in the double-blind treatment period and had evaluable SCORAD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 103 | 107 | 112 | 112
units on a scale | -20.93 (1.894) | -24.82 (1.880) | -26.08 (1.857) | -28.55 (1.867)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.1317, Mixed Models Analysis; LS Mean difference (Final Values) = -3.89, 95% CI 2-sided [-8.95 to 1.17], Standard Error of Mean 2.576
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.0451, Mixed Models Analysis; LS Mean difference (Final Values) = -5.15, 95% CI 2-sided [-10.19 to -0.11], Standard Error of Mean 2.564
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0031, Mixed Models Analysis; LS Mean difference (Final Values) = -7.62, 95% CI 2-sided [-12.66 to -2.58], Standard Error of Mean 2.566

12. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. SCORAD90 is defined as a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 3.3 | 1.7 | 5.0 | 12.5
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.4238, Regression, Logistic; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.11 to 2.49]
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.5118, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.44 to 5.08]
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0129, Regression, Logistic; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.34 to 11.52]

13. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: Body surface area affected by atopic dermatitis will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of atopic dermatitis. LS Means calculated using MMRM model with treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants in the double-blind treatment period and had evaluable BSA data.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 105 | 109 | 113 | 115
percentage of body surface area | -20.31 (1.622) | -21.83 (1.608) | -22.06 (1.581) | -25.66 (1.593)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.4852, Mixed Models Analysis; LS Mean difference (Final Values) = -1.51, 95% CI 2-sided [-5.77 to 2.75], Standard Error of Mean 2.168
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.4205, Mixed Models Analysis; LS Mean difference (Final Values) = -1.74, 95% CI 2-sided [-5.98 to 2.50], Standard Error of Mean 2.160
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0138, Mixed Models Analysis; LS Mean difference (Final Values) = -5.34, 95% CI 2-sided [-9.59 to -1.10], Standard Error of Mean 2.161

14. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment
Time Frame: Week 16
Population: All randomized participants in the double-blind treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
Percentage of participants | 5.7 | 5.0 | 3.3 | 2.5
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.540, Fisher Exact
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.302, Fisher Exact

15. Secondary Outcome: Mean Number of Days Without Use of Background Topical Corticosteroid (TCS)
Description: Mean number of days without use of background TCS was presented. The ANOVA model includes treatment, age cohort, region, and baseline disease severity (IGA) as factors.
Time Frame: Baseline Through 16 Weeks
Population: All randomized participants in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
days | 27.74 (4.06) | 32.22 (4.07) | 30.86 (4.06) | 39.91 (4.10)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.375, ANOVA; LS Mean difference (Final Values) = 4.47, 95% CI 2-sided [-5.41 to 14.35], Standard Error of Mean 5.03
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.536, ANOVA; LS Mean difference (Final Values) = 3.12, 95% CI 2-sided [-6.76 to 13.00], Standard Error of Mean 5.03
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.016, ANOVA; LS Mean difference (Final Values) = 12.17, 95% CI 2-sided [2.29 to 22.05], Standard Error of Mean 5.03

16. Secondary Outcome: Mean Gram Quantity of TCS Use (Tube Weights)
Description: The dispensed TCS tubes were weighed with cap (without the carton) to determine the dispensed amount of TCS in grams. Returned tubes were weighed with cap (without the carton) to determine the amount of TCS in grams used at each visit. Analysis was done via analysis of variance (ANOVA), with geographic region, baseline disease severity, and treatment as factors in the model.
Time Frame: Baseline through 16 Weeks
Population: All randomized participants in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 122 | 121 | 120 | 120
grams | 265.79 (22.04) | 216.60 (22.09) | 228.41 (22.05) | 185.42 (22.26)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.073, ANOVA; LS Mean difference (Final Values) = -49.19, 95% CI 2-sided [-102.81 to 4.42], Standard Error of Mean 27.28
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.172, ANOVA; LS Mean difference (Final Values) = -37.38, 95% CI 2-sided [-91.00 to 16.23], Standard Error of Mean 27.29
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.004, ANOVA; LS Mean difference (Final Values) = -80.37, 95% CI 2-sided [-133.98 to -26.75], Standard Error of Mean 27.28

17. Secondary Outcome: Change From Baseline in Itch NRS for Participants 10 to <18 Years at Study Entry
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LS Means were calculated using mixed model repeated measures (MMRM) model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (10 to <18 years) in the double-blind treatment period and had evaluable Itch NRS data.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 65 | 69 | 78 | 79
units on a scale | -1.15 (0.276) | -1.80 (0.266) | -1.65 (0.261) | -2.25 (0.258)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.0829, Mixed Models Analysis; LS Mean difference (Final Values) = -0.65, 95% CI 2-sided [-1.38 to 0.08], Standard Error of Mean 0.372
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.1752, Mixed Models Analysis; LS Mean difference (Final Values) = -0.50, 95% CI 2-sided [-1.22 to 0.22], Standard Error of Mean 0.368
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0029, Mixed Models Analysis; LS Mean difference (Final Values) = -1.10, 95% CI 2-sided [-1.82 to -0.38], Standard Error of Mean 0.366

18. Secondary Outcome: Change From Baseline in the Parent-Reported Itch Severity Measure (PRISM) for Participants 2 to <10 Years at Study Entry
Description: The Parent-Reported Itch Severity Measure (PRISM) is a single-item, parent/caregiver administered scale that reports the overall severity of their child's itching. Parent/Caregiver's report the overall severity of their child's itching based on observed actions of the child in the past 24 hours. Response options range include "No Itch," "Mild," "Moderate," "Severe," and "Very Severe." The PRISM will be completed for participants <10 years old by the parent/caregiver.
  LS Means were calculated using mixed model repeated measures (MMRM) model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (2 to <10 years old) in the double-blind treatment period and had evaluable PRISM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo Double-blind: Participants 2 to < 10 years received placebo as oral suspension.
- Baricitinib Double-blind Low Dose: Participants 2 to < 10 years received Baricitinib low dose (0.5 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
- Baricitinib Double-blind Medium Dose: Participants 2 to < 10 years received Baricitinib medium dose (1 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
- Baricitinib Double-blind High Dose: Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 31 | 29 | 27 | 21
units on a scale | -0.02 (0.139) | -0.24 (0.146) | -0.49 (0.145) | -0.37 (0.158)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.2688, Mixed Models Analysis; LS Mean difference (Final Values) = -0.21, 95% CI 2-sided [-0.60 to 0.17], Standard Error of Mean 0.193
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.0166, Mixed Models Analysis; LS Mean difference (Final Values) = -0.47, 95% CI 2-sided [-0.85 to -0.09], Standard Error of Mean 0.193
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0908, Mixed Models Analysis; LS Mean difference (Final Values) = -0.34, 95% CI 2-sided [-0.75 to 0.06], Standard Error of Mean 0.202

19. Secondary Outcome: Change From Baseline on the Patient-Oriented Eczema Measure (POEM) Total Score
Description: The POEM is a simple, 7-item, patient-administered scale that assesses disease severity in children and adults. Participants respond to questions about the frequency of 7 symptoms (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) over the last week on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). Scores range from 0-28 with higher total scores indicating greater disease severity.
  LS Means were calculated using MMRM model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants in the double-blind treatment period and had evaluable POEM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 104 | 107 | 112 | 112
units on a scale | -3.02 (0.708) | -3.93 (0.704) | -4.58 (0.696) | -4.58 (0.702)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.3409, Mixed Models Analysis; LS Mean difference (Final Values) = -0.91, 95% CI 2-sided [-2.79 to 0.97], Standard Error of Mean 0.956
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.1022, Mixed Models Analysis; LS Mean difference (Final Values) = -1.56, 95% CI 2-sided [-3.43 to 0.31], Standard Error of Mean 0.952
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.1024, Mixed Models Analysis; LS Mean difference (Final Values) = -1.56, 95% CI 2-sided [-3.43 to 0.31], Standard Error of Mean 0.953

20. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity-Atopic Dermatitis (PGI-S-AD) Score for Participants 10 to <18 Years at Study Entry
Description: The PGI-S-AD is a single-item question asked to the participants on how they would rate their overall atopic dermatitis symptoms over the past 24 hours to evaluate the severity of the disease at that point in time. The 5 categories of responses range from "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe".
  LS Means were calculated using mixed model repeated measures (MMRM) model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (10 to <18 years old) in the double-blind treatment period and had evaluable PGI-S-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 65 | 68 | 78 | 79
units on a scale | -0.33 (0.115) | -0.56 (0.112) | -0.64 (0.109) | -0.83 (0.108)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.1436, Mixed Models Analysis; LS Mean difference (Final Values) = -0.23, 95% CI 2-sided [-0.54 to 0.08], Standard Error of Mean 0.157
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.0483, Mixed Models Analysis; LS Mean difference (Final Values) = -0.31, 95% CI 2-sided [-0.61 to -0.00], Standard Error of Mean 0.154
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0012, Mixed Models Analysis; LS Mean difference (Final Values) = -0.50, 95% CI 2-sided [-0.80 to -0.20], Standard Error of Mean 0.154

21. Secondary Outcome: Change From Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) - Pediatric Depression for Participants 5 to <18 Years at Study Entry
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental and social health in adults and children. The PROMIS Depression item bank assesses self-reported negative mood (sadness, guilt), views on self (self-criticism, worthlessness), social cognition (loneliness, interpersonal alienation), decreased positive affect and engagement (loss of interest, meaning, and purpose). The PROMIS Depression Short Form (8a v2.0 and 6a v2.0) is available in pediatric self-report (ages 8 to <18 years) and for parents/caregivers serving as proxy reporters for children (ages 5 to <8 years). Children aged <5 years will not complete assessment. Both pediatric self-report and proxy-report versions assess depression "in past seven days." Response options range from 1 = Never;2 = Rarely;3 = Sometimes;4 = Often; to 5 = Almost always. Total raw scores were converted to T-Scores (mean= 50 and a standard deviation = 10) with higher scores representing greater depression.
Time Frame: Baseline, Week 16
Population: All randomized participants (5 to <18 years old) in the double-blind treatment period and had evaluable (PROMIS) - Pediatric Depression data. LS Means were calculated using MMRM model, which includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline-by-visit-interaction as fixed continuous effects.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 93 | 102 | 106 | 107
T-score
  5 to <8 years old: number analyzed (Participants) | 11 | 17 | 10 | 18
  5 to <8 years old | -3.95 (2.629) | -2.54 (2.138) | -7.07 (2.644) | -2.83 (2.033)
  8 to <18 years old: number analyzed (Participants) | 82 | 85 | 96 | 89
  8 to <18 years old | -3.60 (1.190) | -3.42 (1.343) | -4.68 (1.034) | -5.30 (1.436)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; for 8 to <18 years old; Test type: Superiority; p = 0.9183, Mixed Models Analysis; LS Mean difference (Final Values) = 0.18, 95% CI 2-sided [-3.27 to 3.63], Standard Error of Mean 1.755
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; for 8 to <18 years old; Test type: Superiority; p = 0.4805, Mixed Models Analysis; LS Mean difference (Final Values) = -1.08, 95% CI 2-sided [-4.09 to 1.93], Standard Error of Mean 1.529
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; for 8 to <18 years old; Test type: Superiority; p = 0.3488, Mixed Models Analysis; LS Mean difference (Final Values) = -1.70, 95% CI 2-sided [-5.26 to 1.86], Standard Error of Mean 1.812
Statistical Analysis 4: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; for 5 to <8 years old; Test type: Superiority; p = 0.2388, Mixed Models Analysis; LS Mean difference (Final Values) = 1.40, 95% CI 2-sided [-4.85 to 7.66], Standard Error of Mean 3.120
Statistical Analysis 5: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; for 5 to <8 years old; Test type: Superiority; p = 0.0098, Mixed Models Analysis; LS Mean difference (Final Values) = -3.13, 95% CI 2-sided [-10.23 to 3.98], Standard Error of Mean 3.542
Statistical Analysis 6: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; for 5 to <8 years old; Test type: Superiority; p = 0.1698, Mixed Models Analysis; LS Mean difference (Final Values) = 1.12, 95% CI 2-sided [-5.18 to 7.42], Standard Error of Mean 3.140

22. Secondary Outcome: Change From Baseline in the PROMIS-Pediatric Anxiety for Participants 5 to <18 Years at Study Entry
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS Anxiety item bank assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). The PROMIS Anxiety Short Form (8 questions, 8a v2.0) is available in a pediatric self-report (ages 8 to <18 years) and for parents/caregivers serving as proxy reporters for their children (youth ages 5 to <8 years old). Children aged <5 years will not complete this assessment. Both pediatric self-report and proxy-report versions assess anxiety "in the past seven days." Response options range from 1= Never; 2 = Rarely; 3 = Sometimes; 4 = Often; to 5 = Almost always. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater anxiety.
Time Frame: Baseline, Week 16
Population: All randomized participants (5 to <18 years old) in the double-blind treatment period and had evaluable (PROMIS) - Pediatric Anxiety data. LS Means were calculated using the MMRM model, which includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline-by-visit-interaction as fixed continuous effects.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 93 | 102 | 106 | 107
T-score
  5 to <8 years old: number analyzed (Participants) | 11 | 17 | 10 | 18
  5 to <8 years old | -4.65 (2.864) | -3.03 (2.318) | -5.09 (2.931) | -3.15 (2.214)
  8 to <18 years old: number analyzed (Participants) | 82 | 85 | 96 | 89
  8 to <18 years old | -4.40 (1.223) | -4.09 (1.394) | -5.44 (1.064) | -6.81 (1.486)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; for 8 to <18 years old; Test type: Superiority; p = 0.8611, Mixed Models Analysis; LS Mean difference (Final Values) = 0.32, 95% CI 2-sided [-3.24 to 3.88], Standard Error of Mean 1.813
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; for 8 to <18 years old; Test type: Superiority; p = 0.5098, Mixed Models Analysis; LS Mean difference (Final Values) = -1.04, 95% CI 2-sided [-4.12 to 2.05], Standard Error of Mean 1.571
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; for 8 to <18 years old; Test type: Superiority; p = 0.1997, Mixed Models Analysis; LS Mean difference (Final Values) = -2.40, 95% CI 2-sided [-6.08 to 1.27], Standard Error of Mean 1.870
Statistical Analysis 4: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; for 5 to <8 years old; Test type: Superiority; p = 0.1957, Mixed Models Analysis; LS Mean difference (Final Values) = 1.62, 95% CI 2-sided [-5.11 to 8.35], Standard Error of Mean 3.351
Statistical Analysis 5: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; for 5 to <8 years old; Test type: Superiority; p = 0.0881, Mixed Models Analysis; LS Mean difference (Final Values) = -0.44, 95% CI 2-sided [-8.19 to 7.32], Standard Error of Mean 3.864
Statistical Analysis 6: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; for 5 to <8 years old; Test type: Superiority; p = 0.1604, Mixed Models Analysis; LS Mean difference (Final Values) = 1.51, 95% CI 2-sided [-5.27 to 8.28], Standard Error of Mean 3.379

23. Secondary Outcome: Change From Baseline in the Children's Dermatology Life Quality Index (CDLQI) at Week 16 for Participants 4 to <18 Years at Study Entry
Description: CDLQI is a validated 10 question tool to measure impact of skin disease on QOL in children by assessing how much the skin problem has affected the subjects over past week. Nine questions were scored as follows: Very much = 3, Quite a lot = 2, Only a little = 1, Not at all or unanswered = 0. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question (max. = 30, min. = 0). Higher the score, the greater the impact on QOL. A negative change from baseline indicated improvement. LS Means were calculated using mixed model repeated measures (MMRM) model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (4 to <18 years old) in the double-blind treatment period and had evaluable CDLQI data.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 97 | 105 | 111 | 111
Score on a Scale | -3.06 (0.480) | -3.73 (0.465) | -3.70 (0.451) | -3.36 (0.459)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.2987, Mixed Models Analysis; LS Mean difference (Final Values) = -0.67, 95% CI 2-sided [-1.93 to 0.59], Standard Error of Mean 0.647
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.3096, Mixed Models Analysis; LS Mean difference (Final Values) = -0.64, 95% CI 2-sided [-1.88 to 0.60], Standard Error of Mean 0.632
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.6341, Mixed Models Analysis; LS Mean difference (Final Values) = -0.30, 95% CI 2-sided [-1.55 to 0.95], Standard Error of Mean 0.635

24. Secondary Outcome: Change From Baseline in Infants' Dermatology Quality of Life Index (IDQOL) at Week 16 for Participants 2 to <4 Years at Study Entry
Description: Infants' Dermatitis Quality of Life Index (IDQOL) is used to evaluate quality of life for subjects of age less than 4 years. IDQOL questionnaires were designed for infants (below the age of 4 years) with atopic dermatitis. The IDQOL was calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score in each questionnaire, the more quality of life is impaired. A negative change from baseline indicated improvement. LS Means were calculated using mixed model repeated measures (MMRM) model includes treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Week 16
Population: All randomized participants (2 to <4 years old) in the double-blind treatment period and had evaluable IDQOL data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 5 | 2 | 1 | 1
units on a scale | -1.40 (1.743) | 3.87 (4.423) | 3.33 (3.752) | -6.40 (3.601)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.2871, Mixed Models Analysis; LS Mean difference (Final Values) = 5.27, 95% CI 2-sided [-6.54 to 17.09], Standard Error of Mean 4.323
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.3093, Mixed Models Analysis; LS Mean difference (Final Values) = 4.73, 95% CI 2-sided [-7.83 to 17.29], Standard Error of Mean 3.835
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.2912, Mixed Models Analysis; LS Mean difference (Final Values) = -5.00, 95% CI 2-sided [-18.22 to 8.21], Standard Error of Mean 3.788

25. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment: Atopic Dermatitis - Caregiver (WPAI-AD-CG) Score
Description: The Atopic Dermatitis Caregiver (WPAI-AD-CG) assesses the effect of a child's atopic dermatitis on the parent/caregiver's work productivity during the past 7 days. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, Scores are calculated as impairment percentages with higher scores indicating greater impairment and less productivity.
  LS Mean were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants in the double-blind treatment period and who had at least 1 post-baseline WPAI measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 96 | 104 | 106 | 109
score on a scale
  Absenteeism: number analyzed (Participants) | 49 | 66 | 62 | 55
  Absenteeism | 3.99 (2.367) | 2.39 (2.135) | 2.14 (2.107) | -0.94 (2.387)
  Presenteeism: number analyzed (Participants) | 55 | 71 | 66 | 59
  Presenteeism | -4.69 (2.719) | -5.62 (2.452) | -9.99 (2.451) | -11.44 (2.797)
  Overall Work Impairment: number analyzed (Participants) | 49 | 66 | 62 | 55
  Overall Work Impairment | 0.38 (3.473) | -3.80 (3.119) | -5.86 (3.086) | -11.15 (3.515)
  Activity Impairment | -7.03 (2.372) | -11.45 (2.318) | -11.90 (2.293) | -14.05 (2.311)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority — Absenteeism Change from Baseline; p = 0.6079, Mixed Models Analysis; LS Mean difference (Final Values) = -1.60, 95% CI 2-sided [-7.74 to 4.54], Standard Error of Mean 3.119
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Absenteeism Change from Baseline; Test type: Superiority; p = 0.5492, Mixed Models Analysis; LS Mean difference (Final Values) = -1.85, 95% CI 2-sided [-7.94 to 4.24], Standard Error of Mean 3.092
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Absenteeism Change from Baseline; Test type: Superiority; p = 0.1338, Mixed Models Analysis; LS Mean difference (Final Values) = -4.93, 95% CI 2-sided [-11.39 to 1.53], Standard Error of Mean 3.281
Statistical Analysis 4: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Presenteeism Change from Baseline; Test type: Superiority; p = 0.7928, Mixed Models Analysis; LS Mean difference (Final Values) = -0.94, 95% CI 2-sided [-7.96 to 6.08], Standard Error of Mean 3.566
Statistical Analysis 5: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Presenteeism Change from Baseline; Test type: Superiority; p = 0.1366, Mixed Models Analysis; LS Mean difference (Final Values) = -5.30, 95% CI 2-sided [-12.30 to 1.69], Standard Error of Mean 3.553
Statistical Analysis 6: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Presenteeism Change from Baseline; Test type: Superiority; p = 0.0760, Mixed Models Analysis; LS Mean difference (Final Values) = -6.75, 95% CI 2-sided [-14.21 to 0.71], Standard Error of Mean 3.792
Statistical Analysis 7: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Overall Work Impairment Change from Baseline; Test type: Superiority; p = 0.3602, Mixed Models Analysis; LS Mean difference (Final Values) = -4.18, 95% CI 2-sided [-13.16 to 4.80], Standard Error of Mean 4.561
Statistical Analysis 8: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Overall Work Impairment Change from Baseline; Test type: Superiority; p = 0.1678, Mixed Models Analysis; LS Mean difference (Final Values) = -6.25, 95% CI 2-sided [-15.14 to 2.65], Standard Error of Mean 4.516
Statistical Analysis 9: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Overall Work Impairment Change from Baseline; Test type: Superiority; p = 0.0170, Mixed Models Analysis; LS Mean difference (Final Values) = -11.54, 95% CI 2-sided [-21.00 to -2.08], Standard Error of Mean 4.808
Statistical Analysis 10: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Activity Impairment Change from Baseline; Test type: Superiority; p = 0.1645, Mixed Models Analysis; LS Mean difference (Final Values) = -4.42, 95% CI 2-sided [-10.66 to 1.82], Standard Error of Mean 3.174
Statistical Analysis 11: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Activity Impairment Change from Baseline; Test type: Superiority; p = 0.1240, Mixed Models Analysis; LS Mean difference (Final Values) = -4.87, 95% CI 2-sided [-11.07 to 1.34], Standard Error of Mean 3.158
Statistical Analysis 12: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Activity Impairment Change from Baseline; Test type: Superiority; p = 0.0270, Mixed Models Analysis; LS Mean difference (Final Values) = -7.02, 95% CI 2-sided [-13.23 to -0.80], Standard Error of Mean 3.163

26. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions-Youth (EQ-5D-Y) for Participants 4 to <18 Years at Study Entry
Description: The EQ-5D-Y questionnaire is health status related and self-completed for pediatric participants ≥8 years old and completed by parents/caregivers for children 4 to <8 years old. Health state profile assessed health in 5 dimensions (Mobility,selfcare,usual activities,pain/discomfort, anxiety/depression) to obtain index score, each with three levels of response (no problems,some problems,a lot of problems). Participants indicated their health state by choosing appropriate level from each dimension. Visual analog scale on which participant rates their perceived health state from 0 ("worst health you can imagine") to 100 ("best health you can imagine") is presented.Higher the score the better the health status. LS Means uses MMRM model which includes treatment,age cohort,region,baseline disease severity(IGA),visit,treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (4 to <18 years old) in the double-blind treatment period with week 16 EQ-5D-Y data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 98 | 105 | 110 | 110
score on a scale | 3.15 (2.090) | 5.12 (2.025) | 5.16 (1.969) | 7.67 (2.000)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.4778, Mixed Models Analysis; LS Mean difference (Final Values) = 1.97, 95% CI 2-sided [-3.49 to 7.43], Standard Error of Mean 2.778
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.4649, Mixed Models Analysis; LS Mean difference (Final Values) = 2.01, 95% CI 2-sided [-3.38 to 7.39], Standard Error of Mean 2.743
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.1013, Mixed Models Analysis; LS Mean difference (Final Values) = 4.52, 95% CI 2-sided [-0.89 to 9.94], Standard Error of Mean 2.755

27. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS) for Participants 10 to <18 Years at Study Entry
Description: Atopic Dermatitis Sleep Scale (ADSS) is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep last night. Item 2, frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times, where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (10 to <18 years old) in the double-blind treatment period with week 16 ADSS Item 2 (frequency of waking) data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 65 | 68 | 78 | 79
score on a scale | -0.42 (0.130) | -0.35 (0.126) | -0.43 (0.123) | -0.55 (0.122)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.6574, Mixed Models Analysis; LS Mean difference (Final Values) = 0.08, 95% CI 2-sided [-0.27 to 0.42], Standard Error of Mean 0.174
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.9488, Mixed Models Analysis; LS Mean difference (Final Values) = -0.01, 95% CI 2-sided [-0.35 to 0.33], Standard Error of Mean 0.172
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.4546, Mixed Models Analysis; LS Mean difference (Final Values) = -0.13, 95% CI 2-sided [-0.47 to 0.21], Standard Error of Mean 0.172

28. Secondary Outcome: Change From Baseline in Skin Pain NRS for Participants 10 to <18 Years at Study Entry
Description: Skin Pain NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours.
  LS Means were calculated using a MMRM model with treatment, age cohort, region, baseline disease severity (IGA), visit, treatment-by-age cohort interaction and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants (10 to <18 years old) in the double-blind treatment period with Week 16 Skin Pain NRS data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Medium Dose | Baricitinib Double-blind High Dose
Number analyzed (Participants) | 65 | 68 | 78 | 79
score on a scale | -1.15 (0.267) | -1.23 (0.259) | -1.56 (0.254) | -1.77 (0.251)
Statistical Analysis 1: Comparison: Placebo Double-blind vs Baricitinib Double-blind Low Dose; Test type: Superiority; p = 0.8133, Mixed Models Analysis; LS Mean difference (Final Values) = -0.09, 95% CI 2-sided [-0.79 to 0.62], Standard Error of Mean 0.360
Statistical Analysis 2: Comparison: Placebo Double-blind vs Baricitinib Double-blind Medium Dose; Test type: Superiority; p = 0.2517, Mixed Models Analysis; LS Mean difference (Final Values) = -0.41, 95% CI 2-sided [-1.11 to 0.29], Standard Error of Mean 0.355
Statistical Analysis 3: Comparison: Placebo Double-blind vs Baricitinib Double-blind High Dose; Test type: Superiority; p = 0.0803, Mixed Models Analysis; LS Mean difference (Final Values) = -0.62, 95% CI 2-sided [-1.32 to 0.08], Standard Error of Mean 0.354

29. Secondary Outcome: Number of Participant Responses With Suspension Acceptability and Palatability Assessment (PK Lead-In) for Participants <10 Years Old at Study Entry
Description: The questionnaire for Suspension acceptability and palatability assessed the participants ability to swallow the oral suspension product, experience relating to the taste, smell and ease of administering and taking the suspension. The questionnaire contained following Questions: Question 1) How did you (your child) like the taste of the medicine? Question 2) How did you (your child) like the smell of the medicine? Question 3) How easy was it for you (your child) to take the medicine today? Question 4) How easy was it for you to use the oral syringe to give your child the dose today? Responses: Liked Very Much, Liked, Neither Liked nor Disliked, Disliked, Disliked Very Much, Very Easy, Easy, Neither Easy nor Hard, Difficult (or Hard) and Very Difficult (or Hard). The number of participants with these responses are presented. Data is presented as "Question Number-Response-Time point".
Time Frame: Week 2
Population: All PK lead-in participants (2 to <10 years old) with data for suspension acceptability and palatability assessment at given time point.
Measure: Number; unit: Participant responses
Groups:
- Baricitinib Open Label High Dose: Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
Arm/Group | Baricitinib Open Label High Dose
Number analyzed (Participants) | 13
Participant responses
  Question 1- Liked Very Much: | 8
  Question 1- Liked | 1
  Question 1- Neither Liked nor Disliked | 3
  Question 1- Disliked | 1
  Question 1- Disliked Very Much | 0
  Question 2- Liked Very Much: | 6
  Question 2- Liked | 1
  Question 2- Neither Liked nor Disliked | 6
  Question 2- Disliked | 0
  Question 2- Disliked Very Much | 0
  Question 3- Very Easy | 8
  Question 3- Easy | 5
  Question 3- Neither Easy nor Hard | 0
  Question 3- Difficult (or Hard) | 0
  Question 3- Very Difficult (or Hard) | 0
  Question 4- Very Easy | 9
  Question 4- Easy | 4
  Question 4- Neither Easy nor Hard | 0
  Question 4- Difficult (or Hard) | 0
  Question 4- Very Difficult (or Hard) | 0

30. Secondary Outcome: Number of Participant Responses With Tablet Acceptability and Palatability Assessment (PK Lead-In) for Participants >=10 Years Old at Study Entry
Description: The questionnaire for tablet acceptability and palatability assessed the participants ability to swallow the tablet. The questionnaire contained the question 1) How easy was it for you (your child) to swallow the medicine today? Responses: Very Easy, Easy, Neither Easy nor Hard, Difficult (or Hard) and Very Difficult (or Hard). The number of participants with these responses are presented. Data is presented as "Question Number-Response-Time point".
Time Frame: Week 2
Population: All PK Lead-In participants >=10 years old, who had data for tablet acceptability and palatability at given time point.
Measure: Number; unit: Participant responses
Groups:
- Baricitinib Open Label High Dose: Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
Arm/Group | Baricitinib Open Label High Dose
Number analyzed (Participants) | 18
Participant responses
  Question 1- Very Easy | 18
  Question 1- Easy | 0
  Question 1- Neither Easy nor Hard | 0
  Question 1- Difficult (or Hard) | 0
  Question 1- Very Difficult (or Hard) | 0

31. Secondary Outcome: Height, Weight and Body Mass Index (BMI) Growth Rate
Description: Height, Weight and BMI Growth Rate will be reported.
Time Frame: 124 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

32. Secondary Outcome: Change of Immunoglobulin G (IgG) Titers
Description: Number of participants with change of IgG titers for tetanus vaccine and pneumococcal conjugate will be presented. A primary immune response was assessed in participants who had never received tetanus or pneumococcal conjugate vaccines previously and secondary/booster responses were assessed if the participants had previously received the vaccines. For pneumococcal conjugate vaccine, number of participants with >= 2-fold increase in >=6 pneumococcal serotypes from pre-vaccination timepoint to specified post-vaccination timepoints through the end of the study will be presented. For tetanus vaccine, number of participants with >= 2-fold increase in participants with baseline titer >=0.1 IU/mL from pre-vaccination timepoint to specified post-vaccination timepoints through the end of the study will be presented.
Time Frame: Baseline Through End of Study Completion
Reporting Status: Not Posted, anticipated posting 2026-05

33. Secondary Outcome: Pop PK: Maximum Observed Drug Concentration at Steady State (Cmax,ss) of LY3009104
Description: Pop PK: Cmax,ss was derived by a population pharmacokinetics approach.
Time Frame: Predose; 0.25 hours (h); 0.5 h; 1 h; 2-4 h; 4 h and 4-6 h post dose
Population: All participants who received at least one dose of study drug in the open-label PK lead-in and double-blind treatment period and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Baricitinib (0.5 mg): Low Dose (2 to<6 Years): Participants 2 to < 6 years of age received Baricitinib low dose (0.5 mg) administered as oral suspension QD.
- Baricitinib (1 mg): Medium Dose (2 to<6 Years): Participants 2 to < 6 years received Baricitinib medium dose (1 mg) administered as oral suspension QD.
- Baricitinib (2 mg): High Dose (2 to<6 Years): Participants 2 to < 6 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Baricitinib (0.5mg): Low Dose (6 to <10 Years): Participants 6 to < 10 years received Baricitinib low dose (0.5 mg) administered as oral suspension QD.
- Baricitinib (1 mg): Medium Dose (6 to <10 Years): Participants 6 to < 10 years received Baricitinib medium dose (1 mg) administered as oral suspension QD.
- Baricitinib (2 mg): High Dose (6 to <10 Years): Participants 6 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
- Baricitinib (1 mg): Low Dose (10 to <18 Years): Participants 10 to < 18 years received Baricitinib low dose (1 mg) administered orally in tablet form QD.
- Baricitinib (2 mg): Medium Dose (10 to <18 Years): Participants 10 to < 18 years received Baricitinib medium dose (2 mg) administered orally in tablet form QD.
- Baricitinib (4 mg): High Dose (10 to <18 Years): Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
Arm/Group | Baricitinib (0.5 mg): Low Dose (2 to<6 Years) | Baricitinib (1 mg): Medium Dose (2 to<6 Years) | Baricitinib (2 mg): High Dose (2 to<6 Years) | Baricitinib (0.5mg): Low Dose (6 to <10 Years) | Baricitinib (1 mg): Medium Dose (6 to <10 Years) | Baricitinib (2 mg): High Dose (6 to <10 Years) | Baricitinib (1 mg): Low Dose (10 to <18 Years) | Baricitinib (2 mg): Medium Dose (10 to <18 Years) | Baricitinib (4 mg): High Dose (10 to <18 Years)
Number analyzed (Participants) | 9 | 8 | 15 | 24 | 26 | 30 | 87 | 86 | 108
nanograms per milliliter (ng/mL) | 18.9 (29) | 35.1 (21) | 64.8 (22) | 11.6 (29) | 23.1 (23) | 44.0 (41) | 13.2 (34) | 27.8 (34) | 50.7 (28)

34. Secondary Outcome: Pop PK: Area Under the Concentration-Time Curve for Dosing Interval at Steady State (AUCtau,ss) of LY3009104
Description: Pop PK: AUCtau,ss was derived by a population pharmacokinetics approach.
Time Frame: Predose; 0.25 hours (h); 0.5 h; 1 h; 2-4 h; 4 h and 4-6 h post dose
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/ mL)
Groups:
- Baricitinib (0.5mg): Low Dose (2 to<6 Years): Participants 2 to < 6 years of age received Baricitinib low dose (0.5 mg) administered as oral suspension QD.
- Baricitinib (4 mg): High Dose (10 to <18years): Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
Arm/Group | Baricitinib (0.5mg): Low Dose (2 to<6 Years) | Baricitinib (1 mg): Medium Dose (2 to<6 Years) | Baricitinib (2 mg): High Dose (2 to<6 Years) | Baricitinib (0.5mg): Low Dose (6 to <10 Years) | Baricitinib (1 mg): Medium Dose (6 to <10 Years) | Baricitinib (2 mg): High Dose (6 to <10 Years) | Baricitinib (1 mg): Low Dose (10 to <18 Years) | Baricitinib (2 mg): Medium Dose (10 to <18 Years) | Baricitinib (4 mg): High Dose (10 to <18years)
Number analyzed (Participants) | 9 | 8 | 15 | 24 | 26 | 30 | 87 | 86 | 108
hour*nanogram per milliliter (h*ng/ mL) | 94.3 (108) | 200 (63) | 298 (51) | 74.8 (64) | 155 (65) | 276 (76) | 109 (63) | 222 (66) | 383 (61)

ADVERSE EVENTS:
Time Frame: Baseline Up to 16 Weeks
Description: All participants who received at least one dose of study drug in the PK Lead-in period (Study period 1) and double-blind treatment period (Study period 2). Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Baricitinib Double-blind Mid Dose: Participants 10 to < 18 years received Baricitinib medium dose (2 mg) and placebo to maintain the blind, administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib medium dose (1 mg) administered as oral suspension QD or placebo oral suspension QD to maintain the blind.
- Baricitinib Open-label High Dose PK Lead-in: Participants 10 to < 18 years received Baricitinib high dose (4 mg) administered orally in tablet form QD.
  Participants 2 to < 10 years received Baricitinib high dose (2 mg) administered as oral suspension QD.
Arm/Group | Placebo Double-blind | Baricitinib Double-blind Low Dose | Baricitinib Double-blind Mid Dose | Baricitinib Double-blind High Dose | Baricitinib Open-label High Dose PK Lead-in
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/120 | 0/120 | 0/120 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/122 | 2/120 | 1/120 | 1/120 | 0/33
Other Adverse Events (participants affected / at risk) | 42/122 | 39/120 | 44/120 | 41/120 | 11/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-blind (N=122) | Baricitinib Double-blind Low Dose (N=120) | Baricitinib Double-blind Mid Dose (N=120) | Baricitinib Double-blind High Dose (N=120) | Baricitinib Open-label High Dose PK Lead-in (N=33)
Corneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Double-blind (N=122) | Baricitinib Double-blind Low Dose (N=120) | Baricitinib Double-blind Mid Dose (N=120) | Baricitinib Double-blind High Dose (N=120) | Baricitinib Open-label High Dose PK Lead-in (N=33)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (3) | 5 (6) | 6 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 3 (3) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 5 (5) | 5 (5) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Impetigo (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4) | 5 (5) | 5 (6) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 4 (4) | 5 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 7 (9) | 11 (20) | 6 (6) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2/64 (3) | 0/62 (0) | 2/63 (5) | 0/53 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 4 (4) | 6 (6) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03952559/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03952559/SAP_001.pdf